CLINICAL TRIAL: NCT00002151
Title: A Randomized, Double-Blind Active-Controlled, Dose-Ranging Study of the Safety and Efficacy of Chronically Administered MDL 28,574A in the Treatment of HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoechst Marion Roussel (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 221C; 028574PR0004; NDPR0004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; AIDS-Related Complex; Zidovudine; MDL 28574
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — celgosivir

INTERVENTIONS:
Drug: Celgosivir hydrochloride

SUMMARY:
To characterize the safety and efficacy of fixed doses of MDL 28,574A administered alone and in combination with zidovudine ( AZT ) in patients with asymptomatic or mildly symptomatic HIV infection. To examine the demographic effects on population pharmacokinetics and pharmacodynamics of MDL 28,574A alone and in combination with AZT.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prior antiretroviral agents for up to 6 months per agent.

Patients must have:

* HIV infection.
* Asymptomatic or mildly symptomatic.
* CD4 count 301 - 500 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following condition are excluded:

Unable or unwilling to comply with study procedures.

Concurrent Medication:

Excluded:

* Chemoprophylactic therapy for mycobacterial infection.
* Any nonstudy prescription medications without approval of investigator.

Patients with the following prior conditions are excluded:

* History of grade 3 or 4 toxicity to <= 600 mg/day AZT.
* History of intolerance to lactose.
* Chronic diarrhea within 6 months prior to study entry.
* Unexplained intermittent or chronic fever, defined as temperature >= 38.5 C for any 7 days within the 30 days prior to study entry.

Prior Medication:

Excluded:

* Antiretroviral therapy within 2 weeks prior to study entry.
* Prior HIV vaccines.
* Biological response modifiers within 30 days prior to study entry.
* Prior foscarnet.
* Any investigational drug with a washout < 5 half-lives prior to study entry.
* Any medications known to alter renal, hepatic, or hematologic / immunologic function (such as barbiturates, phenothiazines, cimetidine, immunomodulators, etc.) within 14 days prior to study entry.

Recent history of alcohol and/or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Clinical Investigations Health Services, Mobile, Alabama
  - California Clinical Trials Med Group, Beverly Hills, California
  - Southwest Community Based AIDS Treatment Group - COMBAT, Los Angeles, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - George Washington Univ / Hershey Med Ctr, Washington D.C., District of Columbia
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - Independent Investigator, Fort Lauderdale, Florida
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Clinical Research Ctr, Sarasota, Florida
  - Independent Investigator, Vero Beach, Florida
  - Ctr for Special Immunology, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - New Orleans Institute of Clinical Investigation, New Orleans, Louisiana
  - Univ Health Ctr, Detroit, Michigan
  - Antibiotic Research Associates, Kansas City, Missouri
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Community Health Network, Rochester, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Infectious Disease Associates, Toledo, Ohio
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Guthrie Clinic, Sayre, Pennsylvania
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Houston Clinical Research Network, Houston, Texas